CLINICAL TRIAL: NCT01506726
Title: A Randomized, Double-Blind, Placebo Controlled Pilot Trial of Oral Salsalate in the Treatment of the Subset of Unexplained Anemia in Elderly Patients With Elevated Interleukin-6
Brief Title: Trial To Evaluate the Efficacy of Oral Salsalate in the Treatment of Older Adults With Unexplained Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug expiration and supply shortage
Sponsor: Harvey Jay Cohen (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Harvey Jay Cohen, Director, Professor and Chair, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00033852; U01AG034661 (NIH)
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Anemia
Keywords: anemia; unexplained anemia; elderly; geriatric; older adults; UAE; over 65; salsalate; PACTTE; pactee; aging; aged; old; older
MeSH Terms: conditions — Anemia | interventions — salicylsalicylic acid; Salicylates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active drug - oral salsalate (Experimental): Subjects randomized to active drug arm will receive 750mg of salsalate (one pill) twice a day (am and pm) for one month. After one month the dose will be increased to 1500mg (2 pills) twice a day (if the 750mg dose was tolerated) for a further 5 months. Total treatment time is 6 months.
  Interventions: Drug: Salsalate
- Placebo Arm (Placebo Comparator): Subjects randomized to the placebo arm will receive a matching placebo pill (one pill) twice a day (am and pm) for one month. After one month the dose will be increased to 2 matching placebo pills twice a day (if the one pill dose was tolerated) for a further 5 months. Total treatment time is 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salsalate — Salsalate 750mg tablet 1 pill bid for one month followed by Salsalate 750mg tablets 2 pills (1500mg) twice a day for a further 5 months (total duration of treatment will be 6 months)
  Other Names: salicylate; salicylate acid
  Arms: Active drug - oral salsalate
Drug: Placebo — Placebo tablet - one pill twice daily for one month, followed by 2 pills twice daily for a further 5 months. Total duration of treatment is 6 months
  Other Names: Placebo tablet
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to determine whether treatment of unexplained anemia in older adults and elevated inflammatory markers with oral salsalate can improve hemoglobin levels and improve physical activity and quality of life.

DETAILED DESCRIPTION:
There is well-defined morbidity and mortality associated with anemia in the elderly and the increasing proportion of elderly adults underscores the population's attributable risk of anemia. As a potentially modifiable factor, an urgent need exists to delineate the impact of anemia correction in the elderly. The Partnership for Anemia: Clinical and Translational Trials in the Elderly (PACTTE) consortium has been created to focus on treatment strategies for anemia in elderly patients. The data presented in this protocol provides a compelling rationale to evaluate the impact of an anti-inflammatory (Salsalate) in older anemic adults with elevated serum iL-6 levels.

Subjects will be 65 years or older adults with unexplained anemia and a elevated serum iL-6 ≥ 1.0 pg/mL.

Subjects will receive 750mg of salsalate or matching placebo (one pill) twice a day (am and pm) for one month. After one month the dose will be increased to 1500mg (2 pills) twice a day (am and pm) if the 750mg dose was tolerated for a further 5 months (for a total of 6 months)

The primary endpoint is to assess whether salsalate improves hemoglobin levels from baseline to 6 month visit.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age 65 years and older, residing in the community or in an assisted-living facility
* Able to adhere to the study visit schedule and other protocol requirements
* Hemoglobin concentration ≥ 9.0 g/dL and < 11.5 g/dL for women and ≥ 9.0 to < 12.7 g/dL for men
* Unexplained anemia (See Appendix 2 for definitions of anemia diagnosis to determine anemia is unexplained)
* Serum IL-6 level ≥ 1.0 pg/mL obtained during screening period (performed at central laboratory).
* Must be able to understand and speak in English; or Spanish speaking subjects who do not speak English may be enrolled per local IRB process and approval, provided the site has appropriate bilingual study staff.

Exclusion Criteria:

* Red blood cell transfusions within the past 3 months
* Estimated glomerular filtration rate (eGFR) of < 30 ml/min (by abbreviated MDRD)
* Use of erythropoiesis stimulating agents (ESA) in the past 3 months
* Active infection defined as symptomatic, requiring active treatment (prophylaxis allowed) or hospitalized for > 24 hours primarily for infection within the past month
* Uncontrolled hypertension defined as diastolic blood pressure > 95 mm Hg or systolic blood pressure > 160 mm Hg on 2 separate occasions during screening period
* Distance on 6MWT above the median for age and sex adjusted population medians (see Table 4)
* Other primary uncorrected cause for anemia including:

  * Known active inflammatory disease including auto-immune diseases (e.g., systemic lupus erythematosis, rheumatoid arthritis, mixed connective tissue disease, sarcoidosis, bronchiolitis obliterans, vasculitis, polymyalgia rheumatica, temporal arteritis, inflammatory bowel disease or related diseases);
  * Chronic active infection (e.g., HIV, viral hepatitis, tuberculosis, osteomyelitis) or receiving therapy within the past 3 months for chronic infection
  * Acute infection within past 3 months (pneumonia, sepsis, bacteremia, prostatitis, urosepsis, pyelonephritis, cholecystitis)
  * Receipt of immunosuppressive therapy in the past 2 years including prednisone except for topical therapy
  * Any cancer (aside from non-melanoma skin cancer) in the past 2 years or on therapy for cancer. In addition, prostate cancer will be excluded if patients have metastatic disease, have had prostatectomy within the prior 6 months, have ever received external beam radiation therapy or brachytherapy, or have received androgen deprivation therapy in the prior 24 months. Subjects with a history of any other form of cancer will likewise be excluded if they have received any radiation or chemotherapy in the prior 24 months.
  * Fecal Occult Blood Test positivity in the past 3 years, Gastrointestinal bleeding in past 3 years and history of peptic ulcer w/ evidence of bleeding
* Elevated AST or ALT ≥ 2x upper limit of normal
* Use of any other experimental drug or therapy within 28 days of initial screening visit
* History of moderate tinnitus affecting instrumental activities of daily activities in the past 3 months
* Current use of acetylsalicylic acid (aspirin) in doses greater than 82 mg/day in the past 3 months. Subjects will also be ineligible if they consume or are expected to consume non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroids, methotrexate, furosemide or anticoagulants during the course of this study.
* Elevated thyroid stimulating hormone (TSH), or other signs of hypothyroid condition. Patients on a stable dose of thyroid replacement are eligible, providing TSH is not elevated.
* Seizure disorder for which phenytoin is used for treatment.
* Hypersensitivity to salsalate, salicylic acid, or acetylsalicylic acid
* History of transient ischemic attacks (TIA), cerebral vascular accident, a clinical diagnosis of angina or myocardial infarction, any coronary interventions (PCI, Bypass, Stent placement) within the prior 12 months to reduce the risk of subject requiring aspirin therapy during the trial
* Dementia defined as the inability to independently provide informed consent and a Montreal Cognitive Assessment (MoCA) score < 22

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Ershler, MD, Principal Investigator — Institute for Advanced Studies in Aging (IASIA); Stanley Schrier, MD, Study Chair — Stanford University; Jeremy Walston, MD, Principal Investigator — Johns Hopkins University
Locations (12):
- United States (12):
  - Lakeview Medical Research, Summerfield, Florida
  - St Joseph's/Candler Health System, Savannah, Georgia
  - University of Illinois, Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Johns Hopkins University Geriatrics Center, Baltimore, Maryland
  - Case Western Reserve University Medical Center, Cleveland, Ohio
  - Clinical Research Solutions, Columbia, Tennessee
  - Clinical Research Solutions, Franklin, Tennessee
  - Clinical Research Solutions, Smyrna, Tennessee
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Institute for Advanced Studies in Aging (IASIA), Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Started | 6 | 5
Completed | 5 | 3
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.2 (3.4) | 74.2 (4.7) | 78.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 3 | 9
  Black or African American | 0 | 1 | 1
  Asian | 0 | 1 | 1
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 11.12 (0.55) | 11.28 (0.34) | 11.19 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin Level From Baseline to 6 Month Visit
Description: To test whether the administration of oral salsalate to a subset of elderly subjects with unexplained anemia (UAE) and high interleukin (IL-6) levels will improve hemoglobin level
Time Frame: baseline; 6 months
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 6 | 5
g/dL | 0.06 (0.76) | 1.00 (0.26)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.230, Wilcoxon (Mann-Whitney); Wilcoxon two sample test; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-2.08 to 0.20]

2. Other Pre Specified Outcome: Change in the 6 Minute Walk Test (6MWT) Distance.
Description: To assess the impact of treatment of anemia with oral salsalate will improve 6 minute walk test (6MWT) distance from baseline to 6 months as measured in meters and centimeters.
Time Frame: baseline; 6 months
Population: Two subjects were missing outcome measure in both the active drug and the placebo arm.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 4 | 3
meters | -20.77 (38.28) | 29.24 (87.99)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.347, t-test, 2 sided

3. Other Pre Specified Outcome: Association Between Change in Hemoglobin and Change in Markers of Inflammation.
Description: To examine whether there is an association between change in hemoglobin and changes in markers of inflammation from prior to study drug to 6 months. Inflammatory markers to be measured are iL-6, Tumor Necrosis Factor alpha Receptor1 (TNF-R1), and C-reactive protein (CRP) in anemia subjects.Correlation between change in the inflammatory markers and the change in HB from prior to study drug to 6 months.
Time Frame: prior to study drug; 6 months
Population: One subject from the active drug oral salsalate group and 2 subjects from the placebo arm group are missing outcomes.
Measure: Number; unit: correlation coefficient
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
correlation coefficient
  IL6 correlation | -0.113 | -0.446
  TNF correlation | 0.948 | -0.977
  CRP correlation | 0.156 | -0.166
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate; Test type: Superiority or Other; p = 0.857, t-test, 2 sided — Correlation between change in IL-6 and change in hemoglobin in the salsalate group. Testing the correlation equal to 0
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority or Other; p = 0.706, t-test, 2 sided — Correlation between change in IL-6 and change in hemoglobin in the placebo group. Testing the correlation equal to 0
Statistical Analysis 3: Comparison: Active Drug - Oral Salsalate; Test type: Superiority or Other; p = 0.014, t-test, 2 sided — Correlation between change in TNF and change in hemoglobin in the salsalate group. Testing the correlation equal to 0
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority or Other; p = 0.136, t-test, 2 sided — Correlation between change in TNF and change in hemoglobin in the placebo group. Testing the correlation equal to 0
Statistical Analysis 5: Comparison: Active Drug - Oral Salsalate; Test type: Superiority or Other; p = 0.803, t-test, 2 sided — Correlation between change in CRP and change in hemoglobin in the salsalate group. Testing the correlation equal to 0
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority or Other; p = 0.894, t-test, 2 sided — Correlation between change in CRP and change in hemoglobin in the placebo group. Testing the correlation equal to 0

4. Secondary Outcome: Change in Markers of Inflammation
Description: To assess whether oral salsalate reduces markers of inflammation including IL-6 and Tumor Necrosis Factor Receptor1 (TNF-R1) in UAE subjects. Change in the marker from prior to study drug to 6 months.
Time Frame: prior to study drug; 6 months
Population: One subject in the active drug oral salsalate group and two subjects in the placebo arm group were missing outcome measures.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
pg/ml
  IL6 | -1.096 (1.210) | 0.703 (1.871)
  Tumor Necrosis Factor Receptor1 (TNF-R1), | 133.48 (390.99) | -189.40 (260.91)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.143, t-test, 2 sided — P value comparing change in IL6 between treatment groups
Statistical Analysis 2: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.257, t-test, 2 sided — P value comparing the change in TNF between treatment groups

5. Secondary Outcome: Assessment of Serum Biomarkers of Erthropoiesis
Description: To assess whether oral salsalate improves serum biomarkers of erythropoiesis by increasing erythropoietin (Epo) in UAE subjects. Change in the Epo from prior to study drug to 6 months.
Time Frame: prior to study drug; 6 months
Population: One subject in the active drug oral salsalate arm and two subjects in the placebo arm are missing outcome measures.
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
mIU/ml | -0.014 (3.237) | -1.540 (2.982)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.535, t-test, 2 sided — P-value comparing the change in EPO between treatment groups

6. Secondary Outcome: Change in Serum Hepcidin Levels
Description: To compare the change in serum hepcidin levels between treatment groups and whether such a change is proportional to the decline in IL-6 levels. Change in the hepcidin from prior to study drug to 6 months. Positive changes represent increases in hepcidin levels and negative changes represent decreases.
Time Frame: prior to study drug; 6 months
Population: One subject in the active drug oral salsalate arm and 3 subjects in the placebo arm are missing outcome measures.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 2
ng/ml | 0.879 (13.378) | 15.462 (10.329)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.232, t-test, 2 sided

7. Secondary Outcome: Change in Cognitive Outcome Measures-Trail Making Test Part B
Description: To quantify the impact of anemia treatment by salsalate on cognitive outcomes based on the Trail Making Test (TMT) Part B as measured by subjects drawing a line from 25 circled numbers to letters in 300 seconds. The change in seconds per completed circle from baseline to month 6.
Time Frame: baseline; 6 months
Population: Two subjects in the active drug oral salsalate group and 3 in the placebo arm group were missing outcome measure.
Measure: Mean (Standard Deviation); unit: second per completed circle
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 4 | 2
second per completed circle | -0.18 (0.68) | 1.23 (0.69)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.076, t-test, 2 sided

8. Secondary Outcome: Change in Frailty Component Related to Fatigue/ Exhaustion
Description: Subjective fatigue/exhaustion: If any of the following three criteria are met, the patient will be classified as frail for fatigue/exhaustion:
  1. "In the past month, on average, have you been feeling unusually tired during the day?" is answered "yes" and indicated as "all of the time" or "most of the time."
  2. "In the past month, on average, have you felt unusually weak?" is answered "yes" and indicated as "all of the time" or "most of the time."
  3. Energy level on a scale of 0 (no energy) to 10 (most energy) reported as ≤ 3. If the subject answers YES to any of the above noted 3 questions, then they are classified as FRAIL.
  The change in frailty for fatigue/ exhaustion is defined as changing from frail at baseline to not frail at month 6 as reported by the subject.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 2 in the placebo arm group were missing outcome measure.
Measure: Number; unit: participants
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
participants | 1 | 0
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p > 0.999, Chi-squared

9. Secondary Outcome: Change in Cognitive Outcome Measures as Determined by Speed of Processing
Description: To quantify the impact of anemia treatment by salsalate on cognitive outcomes based on speed of processing was derived using the z-scores of the following three tests: (1) TMT Part A seconds per completed circle, (2) simple reaction time from the CogState Detection Task, and (3) choice reaction time from the CogState Identification Task. The composite score for a subject at each time point was defined as the mean of the Z-scores for the three tests at the time point. For each subject, the Z-score for each test at time point was derived by subtracting the subject's score at the time point from the overall baseline mean of the test and then dividing by the overall baseline standard deviation of the test. Positive z-scores indicate a better performance compared to the baseline average.The change in the Z-score from baseline to month 6.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 3 in the placebo arm group were missing outcome measure.
Measure: Mean (Standard Deviation); unit: change in Z-Score
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 2
change in Z-Score | 0.29 (0.53) | 1.42 (1.66)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.187, t-test, 2 sided

10. Secondary Outcome: Change in Cognitive Outcome Measures as Determined by Composite Complex Attention/Executive Processing
Description: To quantify the impact of anemia treatment by salsalate on cognitive outcomes based on Complex attention/executive processing was derived using the z-scores of the following three tests: (1) TMT Part B seconds per completed circle, (2) time score from the CogState One Back Task, and (3) accuracy score from the CogState One Back Task. The composite score for a subject at each time point was defined as the mean of the Z-scores for the three tests at the time point. For each subject, the Z-score for each test at time point was derived by subtracting the overall baseline mean of the test from the subject's score at the time point (accuracy score) or by subtracting the subject's score at the time point from the overall baseline mean of the test (TMT and time score) and then dividing by the overall baseline standard deviation of the test. Positive z-scores indicate a better performance compared to the baseline average. The change in the Z-score from baseline to month 6.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 3 in the placebo arm group were missing outcome measure.
Measure: Mean (Standard Deviation); unit: change in Z-Score
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 2
change in Z-Score | 0.71 (0.67) | -0.07 (0.33)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.193, t-test, 2 sided

11. Secondary Outcome: Change in Cognitive Outcome Measures as Determined by Composite Learning and Memory
Description: To quantify the impact of anemia treatment by salsalate on cognitive outcomes based on Learning and memory was derived using the z-scores of the following three tests: (1) CogState ISL immediate recall score (total score from three learning trials), (2) CogState ISL immediate recall score from the first learning trial, and (3) CogState ISL delayed recall scores. The composite score for a subject at each time point was defined as the mean of the Z-scores for the three tests at the time point. For each subject, the Z-score for each test at time point was derived by subtracting the overall baseline mean of the test from the subject's score at the time point and then dividing by the overall baseline standard deviation of the test. Positive z-scores indicate a better performance compared to the baseline average. The change in the Z-score from baseline to month 6.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 3 in the placebo arm group were missing outcome measure.
Measure: Mean (Standard Deviation); unit: change in Z-Score
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 2
change in Z-Score | 0.15 (1.18) | -0.34 (0.71)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.619, t-test, 2 sided

12. Secondary Outcome: Change in Self Reported Outcomes Measures as Reported by Short Form-36 (SF-36) Physical Component Score (PCS)
Description: To quantify the impact of anemia treatment by salsalate on self-reported outcomes measures by change in SF36 physical component score. The SF-36 form identifies self-report physical function and global measure of quality of life and is a multi-purpose, short-form health survey consisting of 36 questions. The Physical Component Summary (PCS) is a subscale of the SF-36 that correlates with physical health domains of the SF-36 ( Physical Function, Role-Physical, and Bodily Pain). The change is calculated and compared from baseline to 6 months. The SF-36 PCS score is a norm based sore with a mean of 50 and standard deviation of 10 where results above and below 50 are above and below the average, respectively, in the 2009 general US population.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 2 in the placebo arm group were missing outcome measure.
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
t score | 1.63 (7.30) | 3.77 (1.38)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.642, t-test, 2 sided

13. Secondary Outcome: Change in Self Reported Outcomes Measures as Reported by FACIT-AN Total Score
Description: To quantify the impact of anemia treatment by salsalate on self -reported outcomes measures by subjects answering 47 questions for patients with anemia and or fatigue. This test detects self-report functional changes and QoL. Change from baseline to 6 months. Scores range from 0-188 with higher scores indicating better function.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 2 in the placebo arm group were missing outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
scores on a scale | 18.9 (19.8) | 7.7 (12.7)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.42, t-test, 2 sided

14. Secondary Outcome: Change in the Frailty Component as Determined by Self-reported Activity Level
Description: To quantify the impact of anemia treatment by salsalate on change in the frailty as measured by change in self-reported activity level. Frailty for activity level is classified by subjects responses to 6physical activity questions on the short version of the Minnesota Leisure Time Activity Questionnaire , were related to walking for exercise, moderately strenuous outdoor chores, dancing, bowling, and regular exercise. The Women's Health And Aging Study (WHAS) scoring algorithm was used to define frailty for self-reported activity level. The answers to these questions were used to calculate kilocalories (Kcals) per week, using the WHAS algorithm, which is further satisfied by by gender. For men, Kcals < 128 per week is frail. For women, Kcals < 90 per week is frail. This is a categorical measurement of yes or no. The outcome is the number of participants who were classified as "frail" at baseline and changed to "not frail" at 6 months.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 2 in the placebo arm group were missing outcome measure.
Measure: Number; unit: participants
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
participants | 1 | 0
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p > 0.999, Chi-squared

15. Secondary Outcome: Change in Frailty Component as Determined by Grip Strength
Description: To quantify the impact of anemia treatment by salsalate on change in the frailty as measured by change in grip strength. Subjects squeeze the grip strength machine 3 times with each hand. For the frailty outcome the maximum grip strength from the dominant hand is used. (change from frail at baseline to not frail at 6 months). Grip strength is stratified by gender and BMI. For men with (BMI <= 24 and a grip strength (GS) <= 29) or (BMI 24.1-28 and grip strength <= 30) or (BMI >28 and a grip strength <= 32) were classified as "frail". For women with (BMI <= 23 and a grip strength of <= 17) or (BMI 23.1-26 and a GS <= 17.3) or (BMI 26.1-29 and a GS <= 18) or (BMI > 29 and a GS <= 21) were classified as "frail".The outcome is the number of participants who were classified as "frail" at baseline and changed to "not frail" at 6 months.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 2 in the placebo arm group were missing outcome measure.
Measure: Number; unit: participants
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
participants | 0 | 1
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.375, Chi-squared

16. Secondary Outcome: Change in Frailty Component as Determined by the 4 Meter Walk Speed
Description: To quantify the impact of anemia treatment by salsalate on change in the speed of the 4 meter walk speed. Subjects are asked to walk as fast as they can for 4 meters. Frailty was determined by the subject's speed. (change from frail at baseline to not frail at 6 months). 4 m walking speed is stratified by gender and height. For men, (height of <= 173 cm and a walking speed of <= 0.65 meter/sec) or a (height > 173, <= .76 meter/sec) were classified as "frail". For women, (height of <= 159 cm and a walking speed of <=.65 meter/sec) or (height >159 cm <= 0.76 meter/sec) were classified as "frail".The outcome is the number of participants who were classified as "frail" at baseline and changed to "not frail" at 6 months.
Time Frame: baseline; 6 months
Population: One subject in the active drug oral salsalate group and 2 in the placebo arm group were missing outcome measure.
Measure: Number; unit: participants
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
participants | 0 | 0

17. Secondary Outcome: Change in Markers of Inflammation
Description: To assess whether oral salsalate reduces C-reactive protein (CRP) in UAE subjects. Change in the CRP from prior to study drug to 6 months.
Time Frame: prior to study drug; 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
ug/ml | -1.976 (1.676) | 1.890 (6.267)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.398, t-test, 2 sided

18. Secondary Outcome: Assessment of Serum Biomarkers of Erthropoiesis
Description: To assess whether oral salsalate improves serum biomarkers of erythropoiesis by decreasing growth differentiation factor-15 (GDF-15) in UAE subjects. Change in the GDF-15 from prior to study drug to 6 months.
Time Frame: prior to study drug; 6 months
Population: One subject in the active drug oral salsalate arm and two subjects in the placebo arm are missing outcome measures.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Number analyzed (Participants) | 5 | 3
pg/ml | 16.688 (308.863) | 187.240 (139.226)
Statistical Analysis 1: Comparison: Active Drug - Oral Salsalate vs Placebo Arm; Test type: Superiority or Other; p = 0.412, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: All non-serious adverse events and serious adverse events will be collected from the time of randomization through the subject's final study visit up to 6 months.
Description: Adverse events and serious adverse events will be collected for subjects who terminate early from the study until the time of their withdrawal.
Arm/Group | Active Drug - Oral Salsalate | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug - Oral Salsalate (N=6) | Placebo Arm (N=5)
Diarrheoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
hypoascusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug - Oral Salsalate (N=6) | Placebo Arm (N=5)
diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
abdominal upper pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
malaise (General disorders) | 0 (0) | 2 (2)
crepitations (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
oedema peripheral (General disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
weight decreased (Investigations) | 0 (0) | 2 (2)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No